CLINICAL TRIAL: NCT05318508
Title: Sagittal Spinopelvic Parameters in Patients With Lower Extremity Amputation
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Assoc. Prof, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E2-21-1002
Record Dates: First submitted 2022-03-28; First posted 2022-04-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Amputation, Traumatic; Low Back Pain
MeSH Terms: conditions — Amputation, Traumatic; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with low back pain
  Interventions: Other: Measurements of sagittal spinopelvic parameters
- patients without low back pain
  Interventions: Other: Measurements of sagittal spinopelvic parameters

INTERVENTIONS:
Other: Measurements of sagittal spinopelvic parameters — Sagittal spinopelvic parameters will be measured from lateral cervicothoracolumbar radiographs of patients with lower extremity amputation.

SUMMARY:
The aim of this study is to investigate the relationship between sagittal spinopelvic parameters and low back pain and quality of life in individuals with lower extremity amputation.

DETAILED DESCRIPTION:
Low back pain is one of the secondary health problems that negatively affect functionality, independence and quality of life in individuals with lower extremity amputation. The prevalence of low back pain was reported to be higher in individuals with lower extremity amputation (52-89%) than in the non-amputee population (12-45%). Although the etiology of low back pain is multifactorial, changing anatomy and biomechanics after lower extremity amputation and maintaining daily activities are often associated with the development of low back pain. Postural imbalance, which is one of the musculoskeletal disorders of the spine that contributes to low back pain, is considered to cause additional load on the spinal structures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 and ≤ 65 years
* Patients followed for at least 12 months with lower extremity amputation
* Patients who have been using prosthesis for at least 3 months
* Patients with stable medical and psychological status
* Patients willing to participate in the study

Exclusion Criteria:

* Patients with serious cardiovascular, pulmonary, neurological disease or other musculoskeletal problems (inflammatory rheumatic disease, active synovitis, severe low back pain, hip/knee joint replacement or other hip/knee-related trauma, fracture, or surgery) that impair walking
* Patients with severe vision, hearing and language problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower extremity amputation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Thoracic kyphosis | baseline
  The angle between the line drawn perpendicular to the line through the T4 upper end plate and the lines drawn perpendicular to the line through the T12 lower end plate.

SECONDARY OUTCOMES:
Cervical lordosis | baseline
Lumbar lordosis | baseline
Pelvic tilt | baseline
Pelvic incidence | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided